CLINICAL TRIAL: NCT05252793
Title: Effect of Education Based on The Health Belief Model on Health Beliefs, Self-Efficacy and Healthy Lifestyle Behaviors in Individuals With Type 2 Diabetes
Brief Title: Effect of Education Based on The Health Belief Model on Healthy Lifestyle Behaviors in Individuals With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sukru Ekenler, Instructor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 178536431
Record Dates: First submitted 2022-02-14; First posted 2022-02-23 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Type 2 Diabetes
Keywords: Self Efficacy; Healthy Lifestyle; Health Belief Model
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Education Program Based on Health Belief Model (Experimental): Experimental: Intervention Patients will be given links to training videos once or twice a week depending on the length of the training module for 6 weeks.
  At the 6th week, the Diabetes Patients Health Belief Model scale, the Diabetes Self-Efficacy Scale and the Healthy Lifestyle Scale-II will be administered as an interim measure.
  Health Belief Model scale in Diabetes Patients, Self-Efficacy Scale in Diabetes and Healthy Lifestyle Scale-II will be applied to the patients at the 12th week as the last measurement.
  Interventions: Behavioral: Education based on the health belief model
- Control (No Intervention): No intervention will be taken against the patients.
  At the 6th week, the Diabetes Patients Health Belief Model scale, the Diabetes Self-Efficacy Scale and the Healthy Lifestyle Scale-II will be administered as an interim measure.
  Health Belief Model scale in Diabetes Patients, Self-Efficacy Scale in Diabetes and Healthy Lifestyle Scale-II will be applied to the patients at the 12th week as the last measurement.

INTERVENTIONS:
Behavioral: Education based on the health belief model — After the intervention, it is expected that the scores of the patients on the healthy lifestyle behaviors scale will increase.
  Arms: Diabetes Education Program Based on Health Belief Model

SUMMARY:
This research will be carried out with a randomized controlled experimental design to examine the effect of education based on the Health Belief Model for individuals with Type 2 Diabetes on their health beliefs, self-efficacy and healthy lifestyle behaviors.

During the research, the relevant polyclinic will be visited regularly. The patients who are followed up in the outpatient clinic for type 2 diabetes will be evaluated in terms of sampling eligibility criteria and their willingness to participate in the research will be questioned. The patients to be included in the study will be randomly assigned to intervention and control groups using the random sampling method. In determining the sample size, two groups, intervention and control, were compared using the "G*Power v3.1.9.4" program. Effect size (d) = 0.80, type I margin of error (α) = 0.05, minimum sample volume to provide test power (1-β) = 0.90, total 68 (experimental group 34, control group 34) is sick. However, it is planned to recruit 20% more patients (41 experiment, 41 control) in order to increase the power and reliability of the research, and there may be losses in the research process.

In the collection of research data; Introductory Characteristics Information Form, Diabetes Health Belief Model Scale, Diabetes Self-Efficacy Scale and Healthy Lifestyle Behaviors Scale-II will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Type 2 Diabetes in the last 6 months
* Being between the ages of 18-65
* HbA1c ≥ 6.0%
* Taking oral antidiabetic medication and/or insulin therapy
* Understanding and speaking Turkish
* Being literate
* Living in Konya
* Not having a communication problem
* Being able to use the WhatsApp® application
* Not having internet access problems
* Individuals who agree to participate in the research by giving their verbal and written consent will be included.

Exclusion Criteria:

* Having a vision problem
* Having mental and communication problems
* Having a neuropsychiatric disorder
* Having a history of malignant disease
* Being pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Healthy Lifestyle Behaviors Scale II Score Change | pre-test (week 1), post-test (week 12)
  Healthy Lifestyle Behaviors Scale II Score Change from Baseline Healthy Lifestyle Behaviors Scale II Score at 12 weeks

SECONDARY OUTCOMES:
Health Belief Model Questionnaire | pre-test (week 1), post-test (week 12)
  Change in perceived severity, perceived susceptibility, perceived benefits, perceived barriers scores at 12 weeks
Self-Efficacy Questionnaire | pre-test (week 1), post-test (week 12)
  Change from Baseline self-efficacy level scores at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sukru EKENLER, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No